CLINICAL TRIAL: NCT06608277
Title: Multi-Center, Randomized, Double-Blind, Placebo-Controlled Trial Comparing Ketamine, Stellate Ganglion Blocks and Combination Treatment to Sham Therapies for Traumatic Brain Injury-Associated Headaches and Post-Traumatic Stress Disorder
Brief Title: Ketamine, SGB and Combination Treatment for TBI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency); Lviv National Medical University (Other); Womack Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Steven Cohen, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00221519
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Posttraumatic Headache; Posttraumatic Stress Disorder
Keywords: Ketamine; Stellate Ganglion Block
MeSH Terms: conditions — Post-Traumatic Headache; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Multi-Center, Randomized, Double-Blind, Placebo-Controlled Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant and outcomes assessor will be blinded to the study group received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A =Stellate ganglion block (SGB) with bupivacaine (LA) plus placebo ketamine (midazolam) (Active Comparator): Stellate ganglion block with the local anesthetic (LA) bupivacaine and placebo (1-7 mg midazolam + normal saline) ketamine.
  The stellate ganglion block will be performed with approximately 8 mL bupivacaine using ultrasound or fluoroscopic guidance. The placebo ketamine will consist of an initial 1-4 mg bolus of midazolam followed by boluses or an infusion (in normal saline) of midazolam up to 7 mg, over 30-60 minutes.
  Interventions: Procedure: Group A active comparator
- Group B = Sham SGB plus ketamine infusion (Active Comparator): Sham SGB will be 1-2 mL of saline given subcutaneously using ultrasound or fluoroscopic guidance. The ketamine will consist of Prior to the sham Stellate Ganglion Block procedure, the study drug ketamine or normal saline will be administered by one of the study team physicians. 100 ml bag will be administered by bolus/infusion or intermittent boluses up to 0.3 mg/kg). The ketamine infusion will start before the sham block where patients will be given 1-4 mg of midazolam + up to 0.3 mg/kg of ketamine, as bolus doses. Over the next 30-60 minutes patients will receive between 0.5-1 mg/kg total dose of ketamine, + additional midazolam as needed.
  Interventions: Drug: Group B active comparator
- Group C = Stellate ganglion block (SGB) with bupivacaine LA plus ketamine infusion (Experimental): These patients will receive both SGB with bupivacaine + ketamine as described above.
  Interventions: Combination Product: Group C Experimental
- Group D = Sham SGB plus placebo ketamine (midazolam) (Placebo Comparator): These patients will receive the sham SGB + placebo ketamine as described above.
  Interventions: Other: Group D Placebo Comparator

INTERVENTIONS:
Procedure: Group A active comparator — Group A placebo comparator. Stellate Ganglion Block plus placebo (.9 normal saline) infusion
  Other Names: Group A
  Arms: Group A =Stellate ganglion block (SGB) with bupivacaine (LA) plus placebo ketamine (midazolam)
Drug: Group B active comparator — Active Comparator: Group B = Sham Stellate Ganglion Block plus ketamine infusion
  Other Names: Group B
  Arms: Group B = Sham SGB plus ketamine infusion
Combination Product: Group C Experimental — Group C experimental Stellate Ganglion Block plus ketamine infusion
  Other Names: Group C
  Arms: Group C = Stellate ganglion block (SGB) with bupivacaine LA plus ketamine infusion
Other: Group D Placebo Comparator — Group D Placebo Comparator: Sham Stellate Ganglion Block plus placebo normal saline
  Other Names: Group D
  Arms: Group D = Sham SGB plus placebo ketamine (midazolam)

SUMMARY:
Post-Traumatic Stress Disorder (PTSD) and traumatic brain injury (TBI) with associated headache are amongst the most common injuries sustained by our deployed forces in Iraq and Afghanistan, as well as in more recent conflicts in Eastern Europe and the Middle East. This study aims to determine whether a procedural intervention (stellate ganglion block (SGB)) or medication (ketamine), alone or in combination, can alleviate PTSD and TBI-associated headache. Determining efficacious treatments in a randomized, double-blind, placebo-controlled, multicenter study trial may improve quality of life in those with TBI and PTSD, and identifying factors associated with treatment outcome (personalized medicine) may enhance selection, thereby improving the risk: benefit and cost-effectiveness ratios.

Primary Objectives:

1. To determine the efficacy of SGB and ketamine infusion as stand-alone treatments for TBI-related headache;
2. To determine the efficacy of SGB and ketamine infusion as stand-alone treatments for PTSD;
3. To determine the comparative effectiveness of SGB and ketamine infusion, and the effect of combination treatment on TBI-related headache and PTSD;
4. Exploratory Aim 1: To determine the effects of SGB, ketamine infusion, and the combination on structural and functional MRI, biomarker levels and pain thresholds and tolerance;
5. Exploratory Aim 2: To identify factors associated with treatment responders overall and for individual treatment groups.

Secondary Objectives:

1. Exploratory Aim 1: To determine the effects of SGB, ketamine infusion, and the combination on structural and functional MRI, biomarker levels and pain thresholds and tolerance (Biomedical levels and MRI not included at Northwestern University Site).
2. Exploratory Aim 2: To identify factors associated with treatment responders overall and for individual treatment groups.

DETAILED DESCRIPTION:
This is a multicenter randomized, double-blind (subject, evaluator) placebo-controlled parallel-group clinical trial where 175 eligible subjects will be randomized into 1 of 4 groups (described below) using a 2:2:2:1 ratio. The purpose of the trial is to test the efficacy and comparative effectiveness of SGB and ketamine infusion on PTSD and post-traumatic headache. There are no reliably effective treatments for either PTSD or TBI-associated headaches, with preliminary and/or conflicting results suggesting efficacy for both SGB and ketamine for both conditions.

The first three groups will receive at least one intervention, with a smaller number receiving sham SGB/ placebo ketamine, which is necessary to determine efficacy and serve as a comparator. Several patient-reported outcomes, including quality of life measures, will be collected at baseline and the primary endpoint at 4 weeks. There will also be patient-reported outcome measures recorded at 1 and 2 weeks. Those with a positive categorical response (described under data collection) at 4 weeks will be followed further at 8 and 12 weeks. Those with negative outcomes will exit the study and be followed as an observational cohort where they will be eligible for non-study measures as determined by the treating providers. This may include other novel treatments such as using higher doses of ketamine, left-sided sympathetic blocks, sympathetic blocks with botulinum toxin and liposomal bupivacaine, and the use of neuromodulation.

For all patients who continue to experience a positive categorical outcome, unblinding will occur at 12 weeks, and they will be followed at 6 months as part of an observational cohort whereby the same outcome measures will be recorded. Those who exit the study and are unblinded at early time points (i.e., 4, 8 or 12 weeks in those with a 12-week negative outcome) will be followed as an observational cohort if they received one of the study treatments, including a variation (e.g., a higher dose of ketamine, a left-sided cervical sympathetic blocks). These time points will be the same as in the clinical trial portion of the study (1,2,4,8 and 12 weeks), and 6 months. For those in either the clinical trial extension or observational cohort who continue to experience a positive outcome at 6 months, we will again follow them at 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years or older
2. Stable doses of medications for > 2 weeks for TBI and/or PTSD
3. For TBI-associated headache with or without PTSD: HIT-6 score of >/=53. For PTSD with or without TBI-associated headache: PCL-5 score >/=33 OR. For those with TBI and PTSD, and a HIT-6 score < 53 and PCL-5 score of <33, individuals with a HIT-6 score of 50-52 and a PCL-5 score of 31 or 32 will be included.
4. Duration of chronic TBI or PTSD > 3 months

Exclusion Criteria:

1. Ketamine infusion or SGB within the past 6 months
2. Serious medical or psychiatric conditions other than TBI or PTSD that could affect cognition (e.g., dementia, Parkinson's Disease)
3. Elevated intracranial pressure
4. For TBI, prior history of headache that can explain the headache intensity (i.e., headache not attributable to TBI)
5. Active psychosis or poorly controlled non-injury or PTSD-related psychiatric condition (e.g., bipolar disorder)
6. Poorly controlled medical conditions that could be exacerbated by treatment (e.g., unstable angina)
7. Pregnancy (women of childbearing age who can become pregnant will have to take a pregnancy test)
8. Non-fluency in English (poor generalizability to military and veteran populations, instruments not validated for use or translated in many languages)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Headache Impact Test (HIT-6) | 4 weeks
  Headache Impact Test (HIT-6) is a 6-item instrument that measures the impact of headaches, scored from 36-78 with higher scores indicating greater disability impact of headaches in a 1-month period that has been validated for a variety of headache conditions, including tension-type headache and migraine.
PTSD Checklist (PCL-5) | 4 weeks
  PTSD Checklist (PCL-5) is a psychometrically-validated 20-item instrument that measures the quality of life in people with posttraumatic stress disorder (PTSD_, scored from 0-80 with higher scores indicating greater disability assesses 20 DSM-5 symptoms of posttraumatic stress disorder.

SECONDARY OUTCOMES:
Central Sensitization Inventory (CSI) | 1 week after procedure
  A 25-item survey which measures central sensitization, scored from 0-100 with higher scores indicating greater sensitization sensitization. It is a self-reported tool that consists of statements related to current health symptoms rated on a 5-point Likert scale, with a score of 40 being the cut off value for central sensitization
Central Sensitization Inventory (CSI) | 2 weeks after procedure
  A 25-item survey which measures central sensitization (amplified nervous system response to sensory stimuli), scored from 0-100 with higher scores indicating greater sensitization sensitization. It is a self-reported tool that consists of statements related to current health symptoms rated on a 5-point Likert scale, with a score of 40 being the cut off value for central sensitization
Central Sensitization Inventory (CSI) | 4 weeks after procedure
  A 25-item survey which measures central sensitization, scored from 0-100 with higher scores indicating greater sensitization sensitization. It is a self-reported tool that consists of statements related to current health symptoms rated on a 5-point Likert scale, with a score of 40 being the cut off value for central sensitization
Central Sensitization Inventory (CSI) | 8 weeks after procedure
  A 25-item survey which measures central sensitization, scored from 0-100 with higher scores indicating greater sensitization sensitization. It is a self-reported tool that consists of statements related to current health symptoms rated on a 5-point Likert scale, with a score of 40 being the cut off value for central sensitization
Central Sensitization Inventory (CSI) | 12 weeks after procedure
  A 25-item survey which measures central sensitization, scored from 0-100 with higher scores indicating greater sensitization sensitization. It is a self-reported tool that consists of statements related to current health symptoms rated on a 5-point Likert scale, with a score of 40 being the cut off value for central sensitization
Headache intensity | 1 week after procedure
  Average and worst headache scores (0-10 numerical rating scale (NRS), overall pain (0=no pain, 10=worst pain imaginable).
  NRS scale)
Headache intensity | 2 weeks after procedure
  Average and worst headache scores (0-10 numerical rating scale (NRS), overall pain (0=no pain, 10=worst pain imaginable).
  NRS scale)
Headache intensity | 4 weeks after procedure
  Average and worst headache scores (0-10 numerical rating scale (NRS), overall pain (0=no pain, 10=worst pain imaginable).
  NRS scale)
Headache intensity | 8 weeks after procedure
  Average and worst headache scores (0-10 numerical rating scale (NRS), overall pain (0=no pain, 10=worst pain imaginable).
  NRS scale)
Headache intensity | 12 weeks after procedure
  Average and worst headache scores (0-10 numerical rating scale (NRS), overall pain (0=no pain, 10=worst pain imaginable).
  NRS scale)
Headache frequency | 1 week after procedure
  Days per week with scores greater or equal to 2, and 7/10 (2= mild headache, 7=severe headache)
Headache frequency | 2 weeks after procedure
  Days per week with scores greater or equal to 2, and 7/10 (2= mild headache, 7=severe headache)
Headache frequency | 4 weeks after procedure
  Days per week with scores greater or equal to 2, and 7/10 (2= mild headache, 7=severe headache)
Headache frequency | 8 weeks after procedure
  Days per week with scores greater or equal to 2, and 7/10 (2= mild headache, 7=severe headache)
Headache frequency | 12 weeks after procedure
  Days per week with scores greater or equal to 2, and 7/10 (2= mild headache, 7=severe headache)
Analgesic or psychotropic medication reduction | 1 week after procedure
  An analgesic or psychotropic medication reduction identified as a > 20% reduction in opioid, barbiturate or benzodiazepine, or cessation of nonopioid analgesic, or > 50% reduction in non-benzodiazepine sedation or psychotropic medication (e.g., antidepressant or antipsychotic).
Analgesic or psychotropic medication reduction | 2 weeks after procedure
  An analgesic or psychotropic medication reduction identified as a > 20% reduction in opioid, barbiturate or benzodiazepine, or cessation of nonopioid analgesic, or > 50% reduction in non-benzodiazepine sedation or psychotropic medication (e.g., antidepressant or antipsychotic).
Analgesic or psychotropic medication reduction | 4 weeks after procedure
  An analgesic or psychotropic medication reduction identified as a > 20% reduction in opioid, barbiturate or benzodiazepine, or cessation of nonopioid analgesic, or > 50% reduction in non-benzodiazepine sedation or psychotropic medication (e.g., antidepressant or antipsychotic).
Analgesic or psychotropic medication reduction | 8 weeks after procedure
  An analgesic or psychotropic medication reduction identified as a > 20% reduction in opioid, barbiturate or benzodiazepine, or cessation of nonopioid analgesic, or > 50% reduction in non-benzodiazepine sedation or psychotropic medication (e.g., antidepressant or antipsychotic).
Analgesic or psychotropic medication reduction | 12 weeks after procedure
  An analgesic or psychotropic medication reduction identified as a > 20% reduction in opioid, barbiturate or benzodiazepine, or cessation of nonopioid analgesic, or > 50% reduction in non-benzodiazepine sedation or psychotropic medication (e.g., antidepressant or antipsychotic).
Headache Impact Test (HIT-6) | 1 week
  Headache Impact Test (HIT-6) is a 6-item instrument that measures the impact of headaches, scored from 36-78 with higher scores indicating greater disability impact of headaches in a 1-month period that has been validated for a variety of headache conditions, including tension-type headache and migraine.
Headache Impact Test (HIT-6) | 2 weeks
  Headache Impact Test (HIT-6) is a 6-item instrument that measures the impact of headaches, scored from 36-78 with higher scores indicating greater disability impact of headaches in a 1-month period that has been validated for a variety of headache conditions, including tension-type headache and migraine.
Headache Impact Test (HIT-6) | 8 weeks
  Headache Impact Test (HIT-6) is a 6-item instrument that measures the impact of headaches, scored from 36-78 with higher scores indicating greater disability impact of headaches in a 1-month period that has been validated for a variety of headache conditions, including tension-type headache and migraine.
Headache Impact Test (HIT-6) | 12 weeks
  Headache Impact Test (HIT-6) is a 6-item instrument that measures the impact of headaches, scored from 36-78 with higher scores indicating greater disability impact of headaches in a 1-month period that has been validated for a variety of headache conditions, including tension-type headache and migraine.
Quality of Life after Brain Injury scale (QoLIBRI) | 1 week
  37-item scale with questions ranging from 1 (not at all) to 5 (very true), with a score ranging from 0-100 (higher numbers indicate better quality of life) calculated from the mean score minus 1, multiplied by 4.
Quality of Life after Brain Injury scale (QoLIBRI) | 2 weeks
  37-item scale with questions ranging from 1 (not at all) to 5 (very true), with a score ranging from 0-100 (higher numbers indicate better quality of life) calculated from the mean score minus 1, multiplied by 4.
Quality of Life after Brain Injury scale (QoLIBRI) | 4 weeks
  37-item scale with questions ranging from 1 (not at all) to 5 (very true), with a score ranging from 0-100 (higher numbers indicate better quality of life) calculated from the mean score minus 1, multiplied by 4.
Quality of Life after Brain Injury scale (QoLIBRI) | 8 weeks
  37-item scale with questions ranging from 1 (not at all) to 5 (very true), with a score ranging from 0-100 (higher numbers indicate better quality of life) calculated from the mean score minus 1, multiplied by 4.
Quality of Life after Brain Injury scale (QoLIBRI) | 12 weeks
  37-item scale with questions ranging from 1 (not at all) to 5 (very true), with a score ranging from 0-100 (higher numbers indicate better quality of life) calculated from the mean score minus 1, multiplied by 4.
Hospital Anxiety and Depression Scale (HADS) | 1 week
  14-item instrument with questions assessing anxiety and depression (7 each) scored from 0-3. For each subscale (anxiety and depression), scores range from 0-21, with higher scores indicating greater pathology.
Hospital Anxiety and Depression Scale (HADS) | 2 weeks after procedure
  Hospital anxiety and depression scale, a 14 question survey scored survey. The anxiety is scored 0 (low) to 21 (high). The depression is scored 0 (low) to 21 (high).
Hospital Anxiety and Depression Scale (HADS) | 4 weeks
  14-item instrument with questions assessing anxiety and depression (7 each) scored from 0-3. For each subscale (anxiety and depression), scores range from 0-21, with higher scores indicating greater pathology.
Hospital Anxiety and Depression Scale (HADS) | 8 weeks
  14-item instrument with questions assessing anxiety and depression (7 each) scored from 0-3. For each subscale (anxiety and depression), scores range from 0-21, with higher scores indicating greater pathology.
Hospital Anxiety and Depression Scale (HADS) | 12 weeks
  14-item instrument with questions assessing anxiety and depression (7 each) scored from 0-3. For each subscale (anxiety and depression), scores range from 0-21, with higher scores indicating greater pathology.
Patient Global Impression of Change Scale | 1 week
  7-item Likert scale with scores ranging from 0 (worse or no change) to 7 (a great deal better)
Patient Global Impression of Change Scale | 2 weeks
  7-item Likert scale with scores ranging from 0 (worse or no change) to 7 (a great deal better)
Patient Global Impression of Change Scale | 4 weeks
  7-item Likert scale with scores ranging from 0 (worse or no change) to 7 (a great deal better)
Patient Global Impression of Change Scale | 8 weeks
  7-item Likert scale with scores ranging from 0 (worse or no change) to 7 (a great deal better)
Patient Global Impression of Change Scale | 12 weeks
  7-item Likert scale with scores ranging from 0 (worse or no change) to 7 (a great deal better)
Positive categorical outcome | 1 week
  Positive is >/= 4 on the PGIC scale and >/= 6-point reduction in HIT-6 and/or a >/= 10-point reduction in PCL-5.
Positive categorical outcome | 2 weeks
  Positive is >/= 4 on the PGIC scale and >/= 6-point reduction in HIT-6 and/or a >/= 10-point reduction in PCL-5.
Positive categorical outcome | 4 weeks
  Positive is >/= 4 on the PGIC scale and >/= 6-point reduction in HIT-6 and/or a >/= 10-point reduction in PCL-5.
Positive categorical outcome | 8 weeks
  Positive is >/= 4 on the PGIC scale and >/= 6-point reduction in HIT-6 and/or a >/= 10-point reduction in PCL-5.
Positive categorical outcome | 12 weeks
  Positive is >/= 4 on the PGIC scale and >/= 6-point reduction in HIT-6 and/or a >/= 10-point reduction in PCL-5.
Sheehan Suicidality Tracking Scale (S-STS) | 4 weeks after procedure
  The S-STS is a short scale designed to assess and monitor suicidality over time and is very sensitive to changes in treatment. The survey has 8 questions with each scored from none (0) to extremely (4).
  outcomes.
International Trauma Questionnaire | 4 weeks
  18-question survey that measures the impact PTSD has on an individual, and helps phenotype PTSD (i.e., into complex PTSD or non-complex). Each question is scored from 0-4 (range 0-72), with higher scores indicating greater disease burden.
International Trauma Questionnaire | 12 weeks
  18-question survey that measures the impact PTSD has on an individual, and helps phenotype PTSD (i.e., into complex PTSD or non-complex). Each question is scored from 0-4 (range 0-72), with higher scores indicating greater disease burden.
PCL-5 | 1 week
  PTSD Checklist (PCL-5) is a psychometrically-validated 20-item instrument that measures the quality of life in people with posttraumatic stress disorder (PTSD_, scored from 0-80 with higher scores indicating greater disability assesses 20 DSM-5 symptoms of posttraumatic stress disorder.
PCL-5 | 2 weeks
  PTSD Checklist (PCL-5) is a psychometrically-validated 20-item instrument that measures the quality of life in people with posttraumatic stress disorder (PTSD_, scored from 0-80 with higher scores indicating greater disability assesses 20 DSM-5 symptoms of posttraumatic stress disorder.
PCL-5 | 8 weeks
  PTSD Checklist (PCL-5) is a psychometrically-validated 20-item instrument that measures the quality of life in people with posttraumatic stress disorder (PTSD_, scored from 0-80 with higher scores indicating greater disability assesses 20 DSM-5 symptoms of posttraumatic stress disorder.
PCL-5 | 12 weeks
  PTSD Checklist (PCL-5) is a psychometrically-validated 20-item instrument that measures the quality of life in people with posttraumatic stress disorder (PTSD_, scored from 0-80 with higher scores indicating greater disability assesses 20 DSM-5 symptoms of posttraumatic stress disorder.
PTSD Checklist (PCL-5) | 1 week
  PTSD Checklist (PCL-5) is a psychometrically-validated 20-item instrument that measures the quality of life in people with posttraumatic stress disorder (PTSD_, scored from 0-80 with higher scores indicating greater disability assesses 20 DSM-5 symptoms of posttraumatic stress disorder.
PTSD Checklist (PCL-5) | 2 weeks
  PTSD Checklist (PCL-5) is a psychometrically-validated 20-item instrument that measures the quality of life in people with posttraumatic stress disorder (PTSD_, scored from 0-80 with higher scores indicating greater disability assesses 20 DSM-5 symptoms of posttraumatic stress disorder.
PTSD Checklist (PCL-5) | 8 weeks
  PTSD Checklist (PCL-5) is a psychometrically-validated 20-item instrument that measures the quality of life in people with posttraumatic stress disorder (PTSD_, scored from 0-80 with higher scores indicating greater disability assesses 20 DSM-5 symptoms of posttraumatic stress disorder.
PTSD Checklist (PCL-5) | 12 weeks
  PTSD Checklist (PCL-5) is a psychometrically-validated 20-item instrument that measures the quality of life in people with posttraumatic stress disorder (PTSD_, scored from 0-80 with higher scores indicating greater disability assesses 20 DSM-5 symptoms of posttraumatic stress disorder.

OTHER OUTCOMES:
Quantitative sensory testing | 4 weeks after procedure
  Quantitative sensory testing will include mechanical temporal summation, a measure of central sensitization, pressure pain thresholds, and the simultaneous presentation of 2 stimuli to assess intrinsic modulation, known as conditioned pain modulation. This test is optional
Serum biomarkers | 4 weeks after procedure
  Markers of inflammation to include interleukins 1 and 6 (IL1 and 6), tumor necrosis factor-alpha (TNF), C-reactive protein (CRP), nerve growth factor (NGF), brain-derived neutrotrophic factor (BDNF), Neurofilament light chain (NfL) and glial fibrillary acidic protein (GFAP). This test is optional.
Structural MRI Imaging | 4 weeks after procedure
  Volumetric changes in gray and white matter, in different regions. This test is optional.
Functional MRI | 4 weeks after procedure
  Functional changes in pain and emotion processing centers (e.g., activation of brainstem, thalamus, hippocampus, insula, anterior cingulate, and somatosensory cortices) as well as changes in connectivity between regions. This test is optional.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Cohen, MD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Anesthesiology Pain Medicine Center, Chicago, Illinois
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Womack Army Medical Center, Fort Bragg, North Carolina